CLINICAL TRIAL: NCT02524197
Title: A Single-Blind, Multiple Ascending-Dose Pilot Study of the Safety, Tolerability, Pharmacokinetics, and Effectiveness of Orally Administered CR845 in Patients With Osteoarthritis of the Hip or Knee
Brief Title: A Study of the Safety and Effectiveness of Orally Administered CR845 in Patients With Osteoarthritis of the Hip or Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR845-CLIN2001-PO
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Osteoarthritis
Keywords: Hip; Knee; Arthritis; pain; CR845; kappa opioid
MeSH Terms: conditions — Osteoarthritis; Arthritis; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- CR845 0.25 mg (Active Comparator): Study medication will be taken b.i.d., in the morning (at least 2 hours before breakfast) and later in the afternoon (at least 2 hours before dinner), beginning on the morning of Day1 at the Baseline Visit.
  Analgesic rescue medication (Acetaminophen) for the treatment of pain will be provided at the Screening Visit.
  Patients will record their daily intake of study medication on the diary provided.
  Interventions: Drug: CR845 0.25 mg
- CR845 0.50 mg (Active Comparator): Study medication will be taken b.i.d., in the morning (at least 2 hours before breakfast) and later in the afternoon (at least 2 hours before dinner), beginning on the morning of Day1 at the Baseline Visit.
  Analgesic rescue medication (Acetaminophen) for the treatment of pain will be provided at the Screening Visit.
  Patients will record their daily intake of study medication on the diary provided.
  Interventions: Drug: CR845 0.50 mg
- CR845 1 mg (Active Comparator): Study medication will be taken b.i.d., in the morning (at least 2 hours before breakfast) and later in the afternoon (at least 2 hours before dinner), beginning on the morning of Day1 at the Baseline Visit.
  Analgesic rescue medication (Acetaminophen) for the treatment of pain will be provided at the Screening Visit.
  Patients will record their daily intake of study medication on the diary provided.
  Interventions: Drug: CR845 1 mg
- CR845 5 mg (Active Comparator): Study medication will be taken b.i.d., in the morning (at least 2 hours before breakfast) and later in the afternoon (at least 2 hours before dinner), beginning on the morning of Day1 at the Baseline Visit.
  Analgesic rescue medication (Acetaminophen) for the treatment of pain will be provided at the Screening Visit.
  Patients will record their daily intake of study medication on the diary provided.
  Interventions: Drug: CR845 5 mg

INTERVENTIONS:
Drug: CR845 0.25 mg — Subjects will dose orally twice a day with CR845 0.25 mg tablets for two weeks. A diary will be kept for recording the individual's pain scores and dosing accountability.
  Arms: CR845 0.25 mg
Drug: CR845 0.50 mg — Subjects will dose orally twice a day with CR845 0.50 mg tablets for two weeks. A diary will be kept for recording the individual's pain scores and dosing accountability.
  Arms: CR845 0.50 mg
Drug: CR845 1 mg — Subjects will dose orally twice a day with CR845 1 mg tablets for two weeks. A diary will be kept for recording the individual's pain scores and dosing accountability.
  Arms: CR845 1 mg
Drug: CR845 5 mg — Subjects will dose orally twice a day with CR845 5 mg tablets for two weeks. A diary will be kept for recording the individual's pain scores and dosing accountability.
  Arms: CR845 5 mg

SUMMARY:
To assess the safety and tolerability of orally-administered CR845 in patients with osteoarthritis (OA) of the hip or knee. The study drug is being tested to reduce OA pain, and will be taken twice a day for two weeks, with four different doses (strengths) being tested. From screening period to follow up examination, the study is expected to last for up to 38 days per participant.

DETAILED DESCRIPTION:
The purpose of this clinical study is to collect information on the effectiveness of CR845 and to look at the safety of different dose levels of CR845 tablets. Oral CR845 has been tested in healthy people. This is the first time that oral CR845 is being tested in patients with osteoarthritis.

Four different doses of CR845 will be tested in this study. Participants will be assigned to one of the four treatment groups. The first 6 participants in each of the 4 treatment groups will be given the study drug in an inpatient study unit (clinic) for approximately 2 days. Frequent blood samples will be taken to measure drug levels during these 2 days. Also, because the study drug (CR845) is known to increase urination during the first day, the amount of fluid that participants drink and the amount of urine that they void during the first day will also be measured.

At the end of the second day, a member of the clinical staff will check vital signs and the patient's laboratory results prior to discharge from the clinic. After that, the remainder of the treatment period is as an outpatient (at home). This involves taking an additional two tablets twice a day, and maintaining a diary that will be returned to the clinic upon completion.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for enrollment if the following criteria are met:

1. Voluntarily provides written informed consent to participate in the study prior to any study procedures.
2. Is able to speak, read, and communicate clearly in English or Spanish; is able to understand the study procedures.
3. Male or female ≥ 25 years of age.
4. BMI ≤ 40
5. Has OA of the hip or knee according to American College of Rheumatology (ACR) criteria.
6. Reports an average pain intensity level ≥ 4 in the index joint at Screening on an NRS.
7. Willing to discontinue currently used pain medications beginning 5 days prior to the Baseline Visit and throughout the study.
8. If female:

   1. Of childbearing potential - the patient must be willing to practice an acceptable form of birth control (defined as the use of an intrauterine device; a barrier method with spermicide; condoms, any form of hormonal contraceptives; or abstinence from sexual intercourse) for the duration of treatment and for at least 3 days following the last dose of study drug.
   2. Of non-childbearing potential - the patient must be surgically or biologically sterile (hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or postmenopausal for at least 1 year).
9. If male, the patient must be surgically or biologically sterile. If not sterile, the patient must agree to use an acceptable form of birth control with a heterosexual partner (as described in inclusion criterion #8) or abstain from sexual relations during the treatment period and for 3 days following the last dose of study drug.
10. Is free of other physical, mental, or medical conditions, which, in the opinion of the Investigator, would make study participation inadvisable.
11. Reports average daily pain intensity ≥ 4 in the index joint during the 3 days prior to Baseline on the NRS.

Exclusion Criteria:

* A patient will be excluded from enrollment if the patient meets any of the following criteria:

  1. Has had a joint replacement in the index joint.
  2. Has received an intra-articular injection of corticosteroids or hyaluronic acid in the index joint within 3 months prior to the Screening Visit.
  3. Has started a new medication for chronic illness within 30 days prior to the Screening Visit.
  4. Has a history or current diagnosis of substance dependence (except caffeine or nicotine) or alcohol abuse, according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
  5. Has a positive urine drug screen for drugs of abuse at Screening or Baseline.
  6. Has been diagnosed with a condition of hyperhidrosis or primary hypodipsia.
  7. Has a history (within 6 months) of clinically meaningful orthostatic changes in vital signs, OR, at Screening, has a decrease in systolic blood pressure by > 20 mm Hg or a decrease in diastolic blood pressure by 10 mm Hg together with an increase in heart rate of > 30 beats per minute when transitioning from supine to standing measurements.
  8. Has a medical condition (e.g., a cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine [adrenal hyperplasia], immunologic, dermatologic, neurologic, oncologic, or psychiatric condition) or a significant laboratory abnormality that, in the Investigator's opinion, would jeopardize the safety of the patient or is likely to confound the study measurements.
  9. Has a serum sodium level > 145 mmol/L at Screening.
  10. Has impaired renal function indicated by serum creatinine > 2 × the reference upper limit of normal (ULN).
  11. Has a serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 × the reference ULN, or total bilirubin > 2 × the ULN at Screening.
  12. Has, in the opinion of the Investigator, any clinical signs of dehydration or hypovolemia (e.g., symptomatic hypotension) or associated laboratory abnormalities (e.g., elevated hematocrit or elevated blood urea nitrogen [BUN] > 1.5 × the reference ULN) at Screening.
  13. Has taken opioid or non-opioid pain medication (e.g., nonsteroidal anti-inflammatory drugs [NSAIDs] such as naproxen or cyclooxygenase-2 inhibitors) within 5 days prior to study drug administration.
  14. Has received another investigational drug within 30 days prior to Baseline or has planned to participate in another clinical trial while enrolled in this study.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To assess the Safety and Tolerability of orally-administered CR845 in patients with osteoarthritis of the hip or the knee, in sequentially escalating doses (0.25 mg, 0.50 mg, 1 mg and 5 mg). | Sentinel cohort initial 48 hours, all subjects 38 days
  The sentinel group will be dosed and monitored in an inpatient clinic unit for 48 hours, then discharged to complete remainder of treatment at home. Following the evaluation of the first group's safety data, the remaining cohorts will begin enrolling. The safety and tolerability of CR845 will be assessed by physical examination, monitoring of adverse events, vital signs, laboratory evaluations, and fluid balance.

SECONDARY OUTCOMES:
To characterize the pharmacokinetic (pk) profile of orally-administered CR845 with twice a day (b.i.d) dosing | 48 hours
  The pharmacokinetic variables for the sentinel groups will have their plasma concentrations summarized and compared to pre-dosing.
To explore the effectiveness of orally administered CR845 in this patient population | 38 days
  The effectiveness of CR845 will be assessed by the measurement of daily joint pain intensity scores (numeric rating scale [NRS]) over time, the impact of treatment on pain, function and stiffness (Western Ontario and McMaster Osteoarthritis Index [WOMAC] and global assessment of OA following treatment (Patient Global Assessment [PGA]).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tiseo, PhD, Study Director — Cara Therapeutics
Locations (5):
- United States (5):
  - Heartland Clinical Research, Omaha, Nebraska
  - Matthew Barton, MD, Las Vegas, Nevada
  - Triad Clinical Trials, LLC, Greensboro, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Investgations of Texas, Plano, Texas